CLINICAL TRIAL: NCT01429987
Title: Study SP304-20210: A Randomized, 12-Week, Double-Blind, Placebo-Controlled, Repeat-Dose, Oral, Dose-Ranging Study to Assess the Safety and Efficacy of Plecanatide in Patients With Chronic Idiopathic Constipation
Brief Title: The Plecanatide Chronic Idiopathic Constipation (CIC) Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP304-20210; SP-SP30420210
Record Dates: First submitted 2011-09-06; First posted 2011-09-07 (Estimated); Results first posted 2017-11-29 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Chronic Idiopathic Constipation
Keywords: Chronic Idiopathic Constipation; Constipation; Sign and Symptoms: Digestive
MeSH Terms: conditions — Constipation | interventions — plecanatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- plecanatide 0.3 mg (Experimental): Subjects receive plecanatide 0.3 mg for 12 consecutive weeks
  Interventions: Drug: plecanatide
- plecanatide 1.0 mg (Experimental): Subjects receive plecanatide 1.0 mg for 12 consecutive weeks
  Interventions: Drug: plecanatide
- plecanatide 3.0 mg (Experimental): Subjects receive plecanatide 3.0 mg for 12 consecutive weeks
  Interventions: Drug: plecanatide
- Placebo (Placebo Comparator): Subjects receive placebo for 12 consecutive weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: plecanatide — Subjects receive experimental study drug for 12 weeks.
  Other Names: Trulance
  Arms: plecanatide 0.3 mg; plecanatide 1.0 mg; plecanatide 3.0 mg
Other: Placebo — Subjects receive experimental study drug for 12 weeks.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo controlled, 12 week repeat oral dose, dose ranging study to determine the efficacy and safety of 3 doses of plecanatide compared to placebo in patients with Chronic Idiopathic Constipation (CIC).

DETAILED DESCRIPTION:
This is a Phase IIb/III, randomized, double-blind, placebo-controlled, 12-Week, Repeat, Oral Dose Ranging, study to determine the safety and efficacy of plecanatide in patients with chronic idiopathic constipation (CIC). Subjects diagnosed with CIC via modified Rome III criteria will be screened against the inclusion and exclusion criteria for the study and enter a 2 Week pre treatment screening. During this phase patients will be required to call in their bowel movements (BM diary) as they occur, and call at least once daily to complete a patient diary of questions on their symptoms (Symptom Diary) associated with CC, as they will throughout the trial. Patients who complete at least 5 days of dosing per week, 6 of each 7 day period of BM diary calls, and continue to have less than 3 complete spontaneous movements per week (as well as meeting other inclusion and exclusion criteria) will be enrolled and randomized to one of three plecanatide doses 0.3 mg, 1.0 mg, and 3.0 mg or placebo. 880 patients will be randomized with the intent of having 200 patients per treatment group (each group the same size) included in efficacy analyses. All subjects receiving at least one dose of plecanatide or matching placebo will be included in the safety analyses.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-75, inclusive
* Body Mass Index = 18-35 kg/m2, inclusive
* Meets modified Rome III criteria for functional chronic idiopathic constipation for at least 3 months with symptom onset for at least 6 months. Note: For this trial, patients with manual maneuvers required for >25% of defecations will not be eligible for participation.
* Less than 3 CSBMs per week at baseline and during pretreatment
* Completed a colonoscopy in accordance with medical guidelines as appropriate, with no clinically significant findings
* Patient is willing to discontinue use of supplemental fiber, laxatives, prescription and nonprescription medications, herbal or dietary supplements intended to treat constipation during the screening, pre-treatment, treatment and 2-week post-treatment periods
* Willing to maintain a stable diet during the study.
* Patients with hemorrhoids and/or diverticulosis (NOT diverticulitis) CAN be entered into the study.

Exclusion Criteria:

* Loose stool (mushy) or watery (Bristol score- 6 or 7) stool in the absence of any laxative or prohibited medicine for > 25% of BMs during the 3 months prior to screening visit OR during the 14 day treatment period
* Patient meets the Rome III criteria for Irritable Bowel Syndrome (IBS-C)
* Active peptic ulcer disease not adequately treated or not stable
* History of cathartic colon, laxative, enema abuse, or ischemic colitis.
* Fecal impaction within 3 months of screening
* Patient has had /has any: diseases or conditions associated with constipation (GI or CNS), structural abnormality of the GI tract or gastric bypass surgery, pelvic floor dysfunction, pseudo-obstruction, active infectious gastritis, diverticulitis, anal fissures or any disease or condition that can affect GI motility or defecation or can be associated with abdominal pain
* Unexplained and clinically significant "alarm symptoms" including lower GI bleeding, iron-deficiency anemia, weight loss or systemic signs of infection or colitis.
* Major surgery within 60 days of screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 951 (Actual)
Dates: Start 2011-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (120):
- United States (120):
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - East Valley Gastroenterology and Hepatology Associates, PC, Chandler, Arizona
  - Genova Clinical Research, Tucson, Arizona
  - Desert Sun Clinical Research, LLC, Tucson, Arizona
  - Adobe Clinical Research, LLC, Tucson, Arizona
  - Preferred Research Partners, Inc, Little Rock, Arkansas
  - ACRI-Phase 1,LLC, Anaheim, California
  - Translational Research Group, INC., d/b/a Providence Clinical Research, Burbank, California
  - GW Research, Inc, Chula Vista, California
  - Community Clinical Trials, Orange, California
  - Dormir Clinical Trials, Inc, Redlands, California
  - Inland Gastroenterology Medical Associates, Inc., Redlands, California
  - Superior Research LLC, Sacramento, California
  - Medical Center for Clinical Research, San Diego, California
  - Medical Associates Research Group, Inc., San Diego, California
  - Progressive Clinical Research, Vista, California
  - Horizons Clinical Research Center, LLC, Denver, Colorado
  - Consultants for Clinical Research of S. Florida, Boynton Beach, Florida
  - Medical Research Unlimited, LLC, Hialeah, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Jupiter Research, Inc., Jupiter, Florida
  - Miami Gastroenterology Consultants, PA, Miami, Florida
  - Advance Medical Research Service Corp, Miami, Florida
  - Advance Medical Research Service, Miami, Florida
  - Florida International Research Center, Miami, Florida
  - Columbus Clinical Services, LLC, Miami, Florida
  - South Medical Research Group, Inc, Miami, Florida
  - Compass Research, LLC, Orlando, Florida
  - Gold Coast Research, LLC, Plantation, Florida
  - DMI Research, Seminole, Florida
  - Meridien Research, Tampa, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Gastro Specialists Research Center, LLC, Decatur, Georgia
  - Mount Vernon Clinical Research, LLC, Sandy Springs, Georgia
  - CTL Research, Eagle, Idaho
  - Advanced Clinical Research, Meridian, Idaho
  - Medex Healthcare Research, Inc., Chicago, Illinois
  - Southwest Gastroenterology Assoc, Oak Lawn, Illinois
  - Rockford Gastroenterology Associates, Ltd., Rockford, Illinois
  - Investigators Research Group, LLC, Brownsburg, Indiana
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Memorial Health System, Inc., d/b/a LaPorte Medical Group, La Porte, Indiana
  - Memorial Health System, Inc., d/b/a Ireland Road Medical Group, South Bend, Indiana
  - Iowa Digestive Disease Center, Clive, Iowa
  - Heartland Research Associates, LLC, Augusta, Kansas
  - Hutchinson Clinic, P.A, Hutchinson, Kansas
  - Heartland Research Associates, LLC, Newton, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Research Integrity, Owensboro, Kentucky
  - Horizon Research Group, LLC, Baton Rouge, Louisiana
  - Gastroenterology Associates, LLC, Baton Rouge, Louisiana
  - Women Under Study, LLC, New Orleans, Louisiana
  - Willis-Knighton Physician Network / Pinnacle Gastroenterology, Shreveport, Louisiana
  - Mid-Atlantic Medical Research Centers, Hollywood, Maryland
  - Boston Clinical Trials, Inc, Boston, Massachusetts
  - NECCR Internal Medicine and Cardiology Associates, LLC, Fall River, Massachusetts
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Beyer Research, Kalamazoo, Michigan
  - Remedica LLC, Rochester, Michigan
  - American Center for Clinical Trials, Southfield, Michigan
  - Ridgeview Research, Chaska, Minnesota
  - The Center for Pharmaceutical Research, PC, Kansas City, Missouri
  - Midwest Center for Clinical Research, Lee's Summit, Missouri
  - St. Louis Center for Clinical Research, St Louis, Missouri
  - Internal Medical Associates of Grand Island, PC, Grand Island, Nebraska
  - Quality Clinical Research Inc., Omaha, Nebraska
  - Central Jersey Medical Research Center, Elizabeth, New Jersey
  - South Jersey Gastroenterology, PA, Marlton, New Jersey
  - Jeffrey Danzig, Ridgewood, New Jersey
  - Albuquerque Clinical Trials, Inc, Albuquerque, New Mexico
  - Lovelace Scientific Resources, Inc, Albuquerque, New Mexico
  - NY Total Medical Care, Brooklyn, New York
  - Synergy First, Brooklyn, New York
  - Long Island Gastrointestinal Research Group LLP, Great Neck, New York
  - Premier Medical Group of the Hudson Valley, PC, Poughkeepsie, New York
  - North American Partners in Pain Management, Valley Stream, New York
  - Paddu and Associates, LLP, Woodside, New York
  - MediSpect, LLC, Boone, North Carolina
  - Clinical and Translational Research Center Hospital, Chapel Hill, North Carolina
  - Carolina Digestive Health Associates, Charlotte, North Carolina
  - Carolina Digestive Health Associates, Davidson, North Carolina
  - LeBauer Research Associates, PA, Greensboro, North Carolina
  - Medoff Medical / Vital re:Search, Greensboro, North Carolina
  - Carolina Digestive Health Associates, Harrisburg, North Carolina
  - Burke Primary Care, Morgantown, North Carolina
  - Wake Research associates, LLC, Raleigh, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Valley Medical Research, Centerville, Ohio
  - Hometown Urgent Care, Columbus, Ohio
  - Hometown Urgent Care and Research, Dayton, Ohio
  - Hometown Urgent Care, Groveport, Ohio
  - Great Lakes Gastroenterology, Mentor, Ohio
  - Hometown Urgent Care and Research, Springfield, Ohio
  - Clinical Research Associates, LLC, Oklahoma City, Oklahoma
  - Consultants in Gastroenerology, Columbia, South Carolina
  - ClinSearch, LLC, Chattanooga, Tennessee
  - Associates in Gastroenterology, Hermitage, Tennessee
  - HCCA Clinical Research Solutions, Jackson, Tennessee
  - PMG Research of Knoxville, Knoxville, Tennessee
  - St. Thomas Medical Group, Nashville, Tennessee
  - KRK Medical Research, Dallas, Texas
  - Research Across America, Dallas, Texas
  - Reasearch Across America, El Paso, Texas
  - Gastroenterology Consultants, Houston, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - Research Across America, Katy, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Digestive Health Center, Pasadena, Texas
  - Quality Research Inc., San Antonio, Texas
  - Spring Gastroenterology PA, Spring, Texas
  - Utah Clinical Trials. LLC, Salt Lake City, Utah
  - Jean Brown Research, Salt Lake City, Utah
  - Advanced Clinical Research, West Jordan, Utah
  - New River Valley Research Institute, Christiansburg, Virginia
  - Clinical Research Partners, LLC, Henrico, Virginia
  - Blue Ridge Medical Research / Gastroenterology Associates of Central Virginia, Lynchburg, Virginia
  - National Clinical Research-Norfolk, Inc, Norfolk, Virginia
  - National Clinical Research-Richmond, Inc., Richmond, Virginia

REFERENCES:
- See also: Sponsor website — http://www.synergypharma.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Plecanatide 0.3 mg: Subjects received plecanatide 0.3 mg orally for 12 consecutive weeks
- Plecanatide 1.0 mg: Subjects received plecanatide 1.0 mg orally for 12 consecutive weeks
- Plecanatide 3.0 mg: Subjects received plecanatide 3.0 mg orally for 12 consecutive weeks
- Placebo: Subjects received placebo orally for 12 consecutive weeks
Period: Overall Study
Arm/Group | Plecanatide 0.3 mg | Plecanatide 1.0 mg | Plecanatide 3.0 mg | Placebo
Started | 238 | 238 | 238 | 237
Completed | 189 | 176 | 202 | 171
Not Completed | 49 | 62 | 36 | 66

BASELINE CHARACTERISTICS:
Population: The mITT population included all randomized patients who received ≥ 1 dose of study drug and ≥ 1 post-baseline BM assessment. 951 patients were randomized; 3 were not treated and 2 received study drug but did not complete a post-dose assessment, yielding 946 patients in the mITT population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Plecanatide 0.3 mg | Plecanatide 1.0 mg | Plecanatide 3.0 mg | Placebo | Total
Number analyzed (Participants) | 237 | 238 | 237 | 234 | 946
Age, Continuous [Mean (Full Range); unit: years] | 47.8 [20 to 75] | 47.1 [18 to 75] | 47.1 [18 to 75] | 46.3 [19 to 75] | 47.1 [18 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 203 | 202 | 205 | 207 | 817
  Male | 34 | 36 | 32 | 27 | 129

OUTCOME MEASURES:

1. Primary Outcome: Overall Responder 9/12 Weeks
Description: A Complete Spontaneous Bowel Movement (CSBM) is a Bowel Movement (BM) that occurs in the absence of laxative use within 24 hours of the BM and the patient reports a feeling of complete evacuation. A weekly responder will have 3 or more CSBMs and an increase of at least one CSBM from baseline in the same week. An overall responder is a patient who is a weekly responder for at least 9 of the 12 treatment weeks, including at least 3 of the last 4 weeks.
Time Frame: 12-Week Treatment Period
Population: The modified Intent-to-Treat (mITT) population is used for all efficacy analyses. The mITT population is all randomized patients who had had at least 1 dose of study drug and who had at least 1 post-baseline BM diary assessment.
Measure: Number; unit: % of Overall Responder 9/12 weeks
Groups:
- Plecanatide 0.3 mg: Subjects received plecanatide 0.3 mg for 12 consecutive weeks
- Plecanatide 1.0 mg: Subjects received plecanatide 1.0 mg for 12 consecutive weeks
- Plecanatide 3.0 mg: Subjects received plecanatide 3.0 mg for 12 consecutive weeks
- Placebo: Subjects received placebo for 12 consecutive weeks
Arm/Group | Plecanatide 0.3 mg | Plecanatide 1.0 mg | Plecanatide 3.0 mg | Placebo
Number analyzed (Participants) | 237 | 238 | 237 | 234
% of Overall Responder 9/12 weeks | 18.6 | 16.8 | 19.0 | 10.7

2. Secondary Outcome: Change From Baseline in 12-week CSBM Weekly Frequency Rate
Description: The number of Complete Spontaneous Bowel Movements (CSBMs) per week
Time Frame: 12-Week Treatment Period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: CSBMs per week
Arm/Group | Plecanatide 0.3 mg | Plecanatide 1.0 mg | Plecanatide 3.0 mg | Placebo
Number analyzed (Participants) | 237 | 238 | 237 | 234
CSBMs per week | 1.60 (0.159) | 1.81 (0.157) | 2.18 (0.159) | 1.09 (0.162)

3. Secondary Outcome: Change From Baseline in 12-week SBM Weekly Frequency Rate
Description: The number of Spontaneous Bowl Movements experienced per week.
Time Frame: 12-Week Treatment Period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: SBMs per week
Arm/Group | Plecanatide 0.3 mg | Plecanatide 1.0 mg | Plecanatide 3.0 mg | Placebo
Number analyzed (Participants) | 237 | 238 | 237 | 234
SBMs per week | 2.20 (0.190) | 2.38 (0.188) | 3.00 (0.191) | 1.35 (0.194)

4. Secondary Outcome: Change From Baseline in Stool Consistency (BSFS) to Over Treatment Period
Description: The stool consistency of each bowel movement (BM) was assessed by patients using the 7-point Bristol Stool Form Scale [BSFS] from 1 to 7.
  1. = separate hard lumps like nuts (difficult to pass)
  2. = sausage shaped but lumpy
  3. = like a sausage but with cracks on its surface
  4. = like a sausage or snake, smooth and soft
  5. = soft blobs with clear-cut edges (passed easily)
  6. = fluffy pieces with ragged edges, a mushy stool
  7. = watery, no solid pieces (entirely liquid)
Time Frame: 12-Week Treatment Period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Plecanatide 0.3 mg | Plecanatide 1.0 mg | Plecanatide 3.0 mg | Placebo
Number analyzed (Participants) | 237 | 238 | 237 | 234
scores on a scale | 1.28 (0.090) | 1.70 (0.090) | 1.97 (0.089) | 0.87 (0.091)

5. Secondary Outcome: Change From Baseline in 12-week Patient Reported Symptoms Associated With Constipation - Straining Score
Description: The severity of straining (Straining Score) was reported by the patients using a 11-point scale (0-10) where 0 = none and 10 = the worst
Time Frame: 12-Week Treatment Period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Plecanatide 0.3 mg | Plecanatide 1.0 mg | Plecanatide 3.0 mg | Placebo
Number analyzed (Participants) | 237 | 238 | 237 | 234
scores on a scale | -1.25 (0.142) | -1.46 (0.142) | -1.73 (0.143) | -1.04 (0.144)

ADVERSE EVENTS:
Description: In the Participate Flow Module-Overall Study, a total of 951 patients were randomized; 3 patients were not treated. Therefore, only 948 treated patients were included in the population at risk. The total number of 948 patients also applied to Other Adverse Events table.
Arm/Group | Plecanatide 0.3 mg | Plecanatide 1.0 mg | Plecanatide 3.0 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/237 | 1/238 | 2/237 | 5/236
Other Adverse Events (participants affected / at risk) | 55/237 | 79/238 | 92/237 | 45/236
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plecanatide 0.3 mg (N=237) | Plecanatide 1.0 mg (N=238) | Plecanatide 3.0 mg (N=237) | Placebo (N=236)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Plecanatide 0.3 mg (N=237) | Plecanatide 1.0 mg (N=238) | Plecanatide 3.0 mg (N=237) | Placebo (N=236)
Diarrhoea (Gastrointestinal disorders) | 13 (13) | 20 (21) | 23 (24) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 6 (6) | 9 (9) | 12 (15) | 11 (11)
Nausea (Gastrointestinal disorders) | 5 (5) | 12 (13) | 8 (8) | 5 (5)
Abdominal Distension (Gastrointestinal disorders) | 5 (5) | 10 (10) | 9 (10) | 5 (5)
Flatulence (Gastrointestinal disorders) | 5 (5) | 3 (3) | 14 (14) | 5 (5)
Urinary Tract Infection (Infections and infestations) | 5 (5) | 9 (10) | 8 (9) | 6 (6)
Upper Respiratory tract infection (Infections and infestations) | 6 (6) | 5 (5) | 9 (10) | 5 (5)
Headache (Nervous system disorders) | 10 (10) | 11 (11) | 9 (9) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes